CLINICAL TRIAL: NCT00656812
Title: Phase II Trial of Rituximab Plus 2CdA in Patients With Advanced or Relapsed Lymphoma of the Mucosa Associated Lymphoid Tissue (MALT)
Brief Title: Rituximab Plus 2CdA in Patients With Advanced or Relapsed Mucosa Associated Lymphoid Tissue (MALT) Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Hoffmann-La Roche (Industry); Lipomed (Industry)
Responsible Party: Prof. Dr. Richard Greil, Arbeitsgemeinschaft medikamentoese Tumortherapie
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_MALT; EudraCT 2008-000767-41
Record Dates: First submitted 2008-04-02; First posted 2008-04-11 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Lymphoma of Mucosa-Associated Lymphoid Tissue
Keywords: advanced MALT lymphoma; Rituximab; 2CdA; chemotherapy; immunotherapy
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): Combination therapy Rituximab plus 2CdA
  Interventions: Drug: Rituximab; Drug: 2-CdA

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 on day 1 of a 21-day treatment cycle
  Other Names: MabThera
Drug: 2-CdA — 0.1 mg/kg s.c. on days 1 - 4 of a 21-day treatment cycle
  Other Names: Litak

SUMMARY:
The purpose of this trial is to evaluate whether a Rituximab plus 2 CdA combination therapy is effective and safe in the treatment of patients with advanced or relapsed lymphoma of the mucosa associated lymphoid tissue (MALT).

DETAILED DESCRIPTION:
Currently, there is no chemotherapeutic standard treatment for patients with MALT lymphoma either presenting with disseminated disease or with relapsing/refractory disease following local treatment (including radiation) or eradication of HP. Various compounds have been tested, including alkylating agents such as cyclophosphamide or chlorambucil, the nucleoside analog cladribine (2CdA), as well as combination regimens including CHOP or MCP (mitoxantrone, chlorambucil, prednisone), but only limited data exists from prospective trials. Thus, trials to evaluate the potential of new compounds in patients with advanced MALT lymphoma are not only justified, but seem warranted.

While systemic approaches were until recently thought to be justified only in patients with disseminated disease, emerging data suggest that also patients with localized disease potentially amenable to radiation may benefit from systemic treatment. This has been demonstrated for ocular adnexal MALT lymphoma and recently also for gastric MALT lymphoma in a randomized fashion, where application of chemotherapy resulted in a significantly longer time to relapse as opposed to surgery or radiation without impairing overall survival.

Both 2CdA and rituximab have been demonstrated as active single agents in MALT lymphoma with mild toxicity profiles and no data on combination therapy with rituximab plus chemotherapy in MALT lymphoma have been published to date. This study will therefore evaluate the efficacy and safety of Rituximab plus 2CdA in patients with advanced or relapsed lymphoma of the mucose associated lymphoid tissue.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of MALT lymphoma of any localization
* Disseminated disease upon diagnosis in case of gastric lymphoma or first or greater relapse after local therapy (including gastrectomy or surgery), prior chemotherapy or HP-eradication. In addition, also patients with localized gastric lymphoma judged refractory to HP-eradication by a minimum follow-up of 12 months after successful HP-eradication can be included in the study.
* Measurable disease
* ECOG performance status of 0,1 or 2
* Age at least 18 years
* Life expectancy of at least 3 months
* Adequate cardiac, renal and liver function tests (LVEF > 50%, serum creatinine < 2.5 mg/dl, ALAT or ASAT < 2.5 x upper limit of normal range (ULN), alkaline phosphatase < 2.5 x ULN, serum bilirubin < 2.0 mg/dl)
* Patient must be willing and able to comply with the protocol for the entire study duration
* Women of child-bearing potential must have a negative pregnancy test and must agree to use effective contraception for the entire treatment period
* Patient's written informed consent

Exclusion Criteria:

* Lymphoma histology other than MALT lymphoma or MALT lymphoma transforming to diffuse large cell lymphoma ("high grade lymphoma")
* Use of any investigational agent 30 days prior to inclusion
* History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the cervix within the last 5 years
* Major surgery, other than diagnostic surgery, within the last 4 weeks
* Evidence of CNS involvement
* A history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months
* Inadequate hematological status at baseline prior to study entry: Dependency on red blood cell and/or platelet transfusions, ANC (absolute neutrophile count (segmented + bands) <1.0 x 109/L
* Patients with active opportunistic infections
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Response rate | After 2, 4 and 6 cycles of therapy

SECONDARY OUTCOMES:
Progression-free survival and relapse-free survival | Duration of study
Occurrence of adverse events | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Markus Raderer, Prof. Dr., Principal Investigator — AKH Wien / Universitaetsklinik fuer Innere Medizin I
Locations (5):
- Austria (5):
  - Universitätsklinikum Graz, Graz
  - Universitaetsklinik Innsbruck/ Klinik für Innere Medizin, Innsbruck
  - Krankenhaus der Stadt Linz, Linz
  - Universitaetsklinik f. Innere Medizin III, Salzburg
  - AKH Wien / Universitaetsklinik fuer Innere Medizin I, Vienna